CLINICAL TRIAL: NCT02061618
Title: Culturally Relevant Exercise for Diabetes (CURE-D)
Acronym: CURE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Principal Investigator, Latha Palaniappan, MD, MS, Associate Investigator, Palo Alto Medical Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-07-250
Record Dates: First submitted 2014-02-10; First posted 2014-02-13 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus
Keywords: South Asian
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention)
- Bollywood Dance Exercise (Experimental): Participants in the Bollywood Dance Exercise group will take part in an 8-week dance intervention. The dance classes will take place 2 times per week, approximately 60 minutes per class, for 8 weeks total.
  Interventions: Behavioral: Bollywood Dance Exercise

INTERVENTIONS:
Behavioral: Bollywood Dance Exercise
  Arms: Bollywood Dance Exercise

SUMMARY:
The Culturally Relevant Exercise for Diabetes (CURE-D) study will determine whether a culturally-sensitive dance intervention is an accepted and effective physical intervention for South Asian women with type 2 diabetes mellitus. The CURE-D study will determine if Bollywood dance exercise improves diabetes outcomes in South Asian women.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Females
* Ethnicity: South Asian
* Hemoglobin A1c ≥ 6.0 mg/dL
* A PAMF patient for ≥ 24 months
* Able and willing to enroll and meet the requirements of the study.

Exclusion Criteria:

* BMI > 35
* Insulin dependent
* Current atrial fibrillation
* Active treatment for cancer
* Diagnosis of a terminal illness and/or in hospice care
* Any serious medical condition which would prevent long-term participation or which would contraindicate physical activity
* Pregnant, lactating, or planning to become pregnant during the study period
* Inability to speak, read, or understand English
* No longer a PAMF patient or planning to transfer care outside of PAMF during the study period
* Investigator discretion for clinical safety or protocol adherence reasons.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Baseline
Hemoglobin A1c | 8-week follow-up
  Change from Baseline in Hemoglobin A1c level at 8 weeks

SECONDARY OUTCOMES:
Body Mass Index | Baseline, 8-week follow-up
Blood Pressure | Baseline, 8-week follow-up
Physical Activity | Baseline, 8-week follow-up
  Assessed by accelerometers

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Medical Foundation Research Institute, Palo Alto, California, United States

REFERENCES:
- [Derived] Natesan A, Nimbal VC, Ivey SL, Wang EJ, Madsen KA, Palaniappan LP. Engaging South Asian women with type 2 diabetes in a culturally relevant exercise intervention: a randomized controlled trial. BMJ Open Diabetes Res Care. 2015 Oct 28;3(1):e000126. doi: 10.1136/bmjdrc-2015-000126. eCollection 2015. PMID 26566446